CLINICAL TRIAL: NCT01873976
Title: Cardiac Biomarkers in Pediatric Cardiomyopathy
Brief Title: Cardiac Biomarkers in Pediatric Cardiomyopathy (PCM Biomarkers)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wayne State University (Other)
Collaborators: Carelon Research (Other); Washington University School of Medicine (Other); Boston Children's Hospital (Other); Columbia University (Other); Children's Hospital of Philadelphia (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Primary Children's Hospital (Other); Monroe Carell Jr. Children's Hospital at Vanderbilt (Other); Stollery Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Montefiore Medical Center (Other); Children's Hospital Colorado (Other); Le Bonheur Children's Hospital (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Steve Lipshultz, Schotanus Family Endowed Chair of Pediatrics, Professor and Chair, Carman and Ann Adams Department of Pediatrics, Wayne State University School of Medicine; President, University Pediatricians and Pediatrician-in-Chief, Children's Hospital of Michigan, Wayne State University
Other Study IDs: 1R01HL109090-01A1 (NIH)
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Incident DCM: A case of dilated cardiomyopathy that presents to the study site for the first time.
- Incident/Recent HCM: A new or existing diagnosis of idiopathic or familial hypertrophic cardiomyopathy, diagnosed within the past 2 months and with a cMRI within 2 months of diagnosis.
- Prevalent HCM or DCM: Any child with a diagnosis of dilated cardiomyopathy or idiopathic or familial hypertrophic cardiomyopathy who has survived transplant-free at least 24 months from the date of cardiomyopathy diagnosis.

SUMMARY:
Cardiomyopathy is a disease of the heart muscle. It is rare, but it can be serious. Cardiomyopathy in children can result in death, disability, heart transplantation or serious heart rhythm disorders. Natural substances in the blood called cardiac biomarkers can be measured in the laboratory and could be a less invasive way (compared to echocardiograms or MRIs) to detect heart dysfunction in children with cardiomyopathy. Little is known about how useful and valid cardiac biomarkers are in the diagnosis and determination of the symptoms in children with cardiomyopathy. The long-term goal of this project is to study how helpful measuring cardiac biomarkers in children with cardiomyopathy is to their doctors in managing the care of these patients as well as improving their overall health. Measures of these cardiac biomarkers could help doctors in determining how best to care for a child with cardiomyopathy, including when to consider heart transplantation as a treatment option.

DETAILED DESCRIPTION:
Pediatric cardiomyopathy is a heterogeneous disease with high morbidity and mortality in which children often present with fulminant disease leading to death or transplant. Highly sensitive and specific cardiac biomarkers or panels of biomarkers, representing different pathologic mechanisms or pathways, are the least invasive (a particularly important consideration in children) and most-cost-effective approach to the early detection of cardiac dysfunction. The long-term goal of this project is to identify such biomarkers in children with cardiomyopathy. These findings could represent a major advance in determining the most appropriate evidence-based clinical care for these children, including when to consider heart transplantation.

The specific aims of this study are:

1. To determine the ability of established and novel cardiac biomarkers to predict short- and long-term outcomes in children with newly diagnosed (incident) dilated cardiomyopathy (DCM)
2. To assess the clinical utility of cardiac biomarkers of collagen metabolism in determining the presence of myocardial fibrosis, as established by cardiac MRI (cMRI), and left ventricular (LV) diastolic dysfunction, as established by echocardiography in both newly diagnosed and existing cases of idiopathic and familial hypertrophic cardiomyopathy (HCM) in children.
3. To determine whether longitudinal changes in cardiac biomarkers are associated with worsening heart failure (HF) class in clinically stable children with dilated or hypertrophic cardiomyopathy. This study will determine the importance of serological biomarkers, in conjunction with cardiac imaging, in the early identification of heart disease before cardiac remodeling and functional impairment have become irreversible in a pediatric population.

This is a 5-year prospective study of up to 480 children with either primary dilated or hypertrophic cardiomyopathy. The study will have three components: 1) clinical data collection by chart review, 2) biospecimen collection and testing, and 3) centralized review and measurement of echocardiograms and cMRIs.

ELIGIBILITY:
Inclusion Criteria:

* Patient is alive and has not received a transplant prior to enrollment in the study.
* Under age 21 years at age of enrollment
* For Group 1 (incident DCM), a case of DCM presenting to a study site within 2 years of the original cardiomyopathy diagnosis
* Group 2 (incident/recent HCM), a new or existing diagnosis of idiopathic or familial HCM with a cMRI within 12 months of diagnosis
* Group 3 (prevalent HCM or DCM), any child with a diagnosis of DCM or idiopathic, familial, or HCM due to a known disease-causing mutation who has survived transplant-free at least 12 months from the date of original cardiomyopathy diagnosis
* For all 3 groups, diagnosis of cardiomyopathy must be confirmed by Echocardiographic or cMRI criteria

Exclusion Criteria:

A patient is not eligible for enrollment if one or more of the following conditions are met at the time of presentation with cardiomyopathy:

* Any cardiomyopathy diagnosis other than DCM or idiopathic HCM, familial HCM or HCM due to a known disease-causing gene
* Endocrine disease known to cause heart muscle disease (including infants of diabetic mothers)
* History of rheumatic fever
* Toxic exposures known to cause heart muscle disease (anthracyclines, mediastinal radiation, iron overload or heavy metal exposure)
* HIV infection or born to an HIV positive mother
* Kawasaki disease
* Congenital heart defects unassociated with malformation syndromes (e.g., valvular heart disease or congenital coronary artery malformations)
* Immunologic disease
* Invasive cardiothoracic procedures or major surgery during the preceding month, except those specifically related to cardiomyopathy including left ventricular assist device (LVAD), extracorporeal membrane oxygenator (ECMO), and automatic implantable cardioverter defibrillator (AICD) placement
* Uremia, active or chronic
* Abnormal ventricular size or function that can be attributed to intense physical training or chronic anemia
* Chronic arrhythmia, unless there are studies documenting inclusion criteria prior to the onset of arrhythmia (except a patient with chronic arrhythmia, subsequently ablated, whose cardiomyopathy persists after two months is not to be excluded)
* Malignancy
* Systemic Hypertension
* Pulmonary parenchymal or vascular disease (e.g., cystic fibrosis, cor pulmonale, or pulmonary hypertension)
* Ischemic coronary vascular disease
* Association with drugs (e.g., growth hormone, corticosteroids, cocaine) or other diseases known to cause hypertrophy

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cases of dilated and hypertrophic cardiomyopathy will be recruited at 11 pediatric cardiology centers in the US and Canada.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Time to Death | 2 years

SECONDARY OUTCOMES:
Time to heart transplant | 2 years
Worsening heart failure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Lipshultz, MD, Principal Investigator — Wayne State University
Locations (13):
- United States (12):
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital of New York, Columbia Presbyterian Medical Center, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UMPC, Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Primary Children's Medical Center, Salt Lake City, Utah
- Stollery Children's Hospital, University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Schmitt W, Diedrich C, Hamza TH, Meyer M, Eissing T, Breitenstein S, Rossano JW, Lipshultz SE. NT-proBNP for Predicting All-Cause Death and Heart Transplant in Children and Adults with Heart Failure. Pediatr Cardiol. 2025 Mar;46(3):694-703. doi: 10.1007/s00246-024-03489-7. Epub 2024 May 9. PMID 38722325
- [Derived] Kirmani S, Woodard PK, Shi L, Hamza TH, Canter CE, Colan SD, Pahl E, Towbin JA, Webber SA, Rossano JW, Everitt MD, Molina KM, Kantor PF, Jefferies JL, Feingold B, Addonizio LJ, Ware SM, Chung WK, Ballweg JA, Lee TM, Bansal N, Razoky H, Czachor J, Lunze FI, Marcus E, Commean P, Wilkinson JD, Lipshultz SE. Cardiac imaging and biomarkers for assessing myocardial fibrosis in children with hypertrophic cardiomyopathy. Am Heart J. 2023 Oct;264:153-162. doi: 10.1016/j.ahj.2023.06.005. Epub 2023 Jun 12. PMID 37315879
- [Derived] Everitt MD, Wilkinson JD, Shi L, Towbin JA, Colan SD, Kantor PF, Canter CE, Webber SA, Hsu DT, Pahl E, Addonizio LJ, Dodd DA, Jefferies JL, Rossano JW, Feingold B, Ware SM, Lee TM, Godown J, Simpson KE, Sleeper LA, Czachor JD, Razoky H, Hill A, Westphal J, Molina KM, Lipshultz SE; Pediatric Cardiomyopathy Registry Investigators. Cardiac Biomarkers in Pediatric Cardiomyopathy: Study Design and Recruitment Results from the Pediatric Cardiomyopathy Registry. Prog Pediatr Cardiol. 2019 Jun;53:1-10. doi: 10.1016/j.ppedcard.2019.02.004. Epub 2019 Mar 7. PMID 31745384